CLINICAL TRIAL: NCT03922074
Title: Outcomes of Colonoscopy With Non-anesthesiologist Administered Propofol. An Equivalence Trial
Brief Title: Outcomes of Colonoscopy With Non-anesthesiologist Administered Propofol
Acronym: ADR_NAAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serveis de Salut Integrats Baix Empordà (Other)
Responsible Party: Principal Investigator, Marco Alburquerque, Head of Gastroenterology Department, Serveis de Salut Integrats Baix Empordà
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 42319_TDA_ANE
Record Dates: First submitted 2019-04-10; First posted 2019-04-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Colo-rectal Cancer; Colon Adenoma; ADR
Keywords: ADR with Non-Anesthesiologist administered propofol (NAAP)
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-anesthesiologist administered propofol (Experimental): Sedation directed by an endoscopist in which the intravenous drugs are propofol and fentanyl . Target level sedation: moderate - deep.
  Interventions: Procedure: Sedation directed by an endoscopist
- Monitored anesthesia care (Active Comparator): Sedation directed by an anesthesiologist in which the used intravenous drugs and target level sedation are chosen by the anesthesiologist.
  Interventions: Procedure: Sedation directed by an anesthesiologist

INTERVENTIONS:
Procedure: Sedation directed by an endoscopist — The nurse begins with fentanyl infusion in bolus: 75 μg (1.5 ml) and initial propofol dose (10mg/ml) in bolus of 0.5 - 2.5 mg/Kg followed by a maintenance dose of 20 - 60ml/h through Target-controlled infusion (TCI) pump. In this way, we get a target level sedation between 1 - 3, according to Observer's Assessment of Alertness/Sedation Scale (OAAS).
  The role of the nurse, directed by an endoscopist, it is exclusively the administration of intravenous drugs and the patient monitorship throughout the procedure.
  Arms: Non-anesthesiologist administered propofol
Procedure: Sedation directed by an anesthesiologist — The choice of the drugs and the target level sedation are directed by an anesthesiologist
  Arms: Monitored anesthesia care

SUMMARY:
The Efficacy and safety of Non-anesthesiologist administered propofol (NAAP) for gastrointestinal endoscopy have been widely documented although there is not information which has evaluated the outcomes of colonoscopy it self when the endoscopist has to fulfill the additional task of supervising the sedation.

Objective: To determine the equivalence of adenoma detection rate (ADR) in colorectal cancer (CRC) screening colonoscopies performed with NAAP and performed with monitored anesthesia care (MAC).

Method: Single blind non-randomized controlled equivalence trial. Patients: Adults between 50 - 69 years old from National CRC screening program (CRCSP). Intervention: The patients are blindly assigned to undergo either colonoscopy with NAAP or MAC according to the arrival of fecal occult blood test, patient's suitability for colonoscopy date and availability of places at endoscopy schedule (with NAAP or MAC).

ELIGIBILITY:
Inclusion Criteria:

Healthy patients -

Exclusion Criteria:

Patients with familial colorectal cancer history

-

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 30 days
  Percentage of patients aged ≥50 years undergoing first-time screening colonoscopy who have one or more conventional adenomas detected and removed